CLINICAL TRIAL: NCT05246410
Title: A Prospective, Multicenter and Randomized Controlled Trial to Evaluate the Efficacy and Safety of a Spot Stent System Using in the Percutaneous Transluminal Angioplasty of Femoropopliteal Arteries.
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of a Spot Stent System Used in Femoropopliteal Arteries.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acoart-08
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Vascular Disease (PVD); Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spot stent system (Experimental): A system that loaded multi low radial force stents on one catheter.
  Interventions: Device: Spot stent system
- Self-Expanding peripheral stent system (Active Comparator): A conventional stent system that commonly used.
  Interventions: Device: Self-expanding peripheral stent system

INTERVENTIONS:
Device: Spot stent system — Spot stent system designed and produced by Acotec
  Arms: Spot stent system
Device: Self-expanding peripheral stent system — Self-expanding peripheral stent system designed and produced by Ev3, Inc
  Arms: Self-Expanding peripheral stent system

SUMMARY:
A prospective randomized trial designed to compare the efficacy and safety of spot stent system versus self-expanding peripheral stent system in the endovascular treatment of femoropopliteal arterial stenotic disease.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to assess the efficacy and safety of spot stent system ,which is indicated for use in patients with atherosclerotic disease of the superficial femoral artery (SFA) or proximal popliteal arteries and for the treatment of insufficient results after percutaneous transluminal angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤80 years old
* Had lower extremity arterial occlusive diseases, and Rutherford classification is 2-5
* Target lesion is in the superficial femoral artery (SFA) and/or proximal popliteal artery (above the knee), located ≥1 cm below the common femoral artery (CFA) bifurcation to the distal segment of the proximal popliteal artery at the superior end of the patella.
* Target lesion had severe stenosis (stenosis degree ≥70%) or occlusion.
* Presence of at least one patent infrapopliteal vessel.
* The length of target lesion ≥10 cm.
* After predilation, the target lesion has <30% residual stenosis and presence of at least one flow-limiting dissection (by visual estimate).
* Subject (or legal guardian) understands the study requirements and procedures and provides written Informed Consent before any study tests or procedures are performed.

Exclusion Criteria:

* The plasma creatinine level is higher than 150 umol/L.
* Thrombolysis or thrombectomy is required.
* The patient had underwent lower-limb arterial surgery or thrombolysis on the target limb within 6 weeks.
* Previously implanted stent in the target lesion.
* The guide wire can not cross the target lesion.
* Angiographic evidence of calcification severe enough that it renders the target lesion non-dilatable.
* Patient has a known allergy to anticoagulant drugs, anti-platelet drugs or contrast medium that cannot be adequately pre-medicated.
* Women who are pregnant or breast-feeding.
* The subjects have participated in other drug property studies or device studies that have not yet completed the main end point.
* Patient has life expectancy of less than 12 months.
* Patient who planned to do above the ankle amputation before the operation.
* Patient who had severe hemorrhage or coagulation disorder which judged by the investigator.
* The investigator think the patient is not suitable for participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary patency rate of target lesion at 12 months post-procedure | 12 months post-procedure
  Defined as freedom from clinically driven target lesion revascularization (CD-TLR) and binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4)

SECONDARY OUTCOMES:
Rate of device success | immediate post-procedure
  Defined as successful delivery, release and retrieval of the device.
Rate of procedural success | 7 days post-procedure
  Defined as no provisional stent implanted or major adverse event occured prior to discharge.
Rate of clinically driven target lesion revascularization within 12 months post-procedure | 12 months post-procedure
  Defined as any reintervention at the target lesion due to the following symptoms: drop of ABI >20% or ABI >0.15 compared to the post-procedure ABI
The change of Rutherford class from baseline | 12 months post-procedure
  Defined as change in target limb Rutherford class from baseline to 12 months
The change of ankle-brachial index (ABI) from baseline | 12 months post-procedure
  Defined as change of target limb ABI from baseline to 12 months
Rate of composite safety endpoint | 30 days post-procedure
  Defined a composite rate of all cause death, major target limb amputation (above-the-ankle amputation), clinically driven target lesion revascularization (CD-TLR) through 30 days post- procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guo Wei, MD, Principal Investigator — Chinese PLA General Hospital
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Zhejiang Provincial People'S Hospital, Zhejiang, Zhejiang